CLINICAL TRIAL: NCT06080308
Title: Research on the Molecular Mechanisms of Liver Ischemia-reperfusion Injury and Clinical Data Analysis: an Observational Study
Brief Title: Liver Ischemia-reperfusion Injury and Clinical Data Analysis
Status: Recruiting | Type: Observational
Sponsor: Qin Zhang (Other)
Responsible Party: Sponsor-Investigator, Qin Zhang, phd, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20230940
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Liver Injury
Keywords: Hepatic ischemia; Reperfusion injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — During the procedure, the remaining blood samples are checked for blood gas analysis, and then plasma is taken
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Searching for new targets for the diagnosis and treatment of liver ischemia-reperfusion injury.

DETAILED DESCRIPTION:
Through the analysis of serological data during liver resection elective surgery with hepatic pedicle occlusion and reperfusion, as well as the analysis of patient-related data, we aim to identify key target points that affect reperfusion injury and explore their underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to participate in the study and has signed an informed consent form. 2) Age ≥ 18 years and ≤ 70 years. 3) ASA classification ≤ III. 4) Criteria for liver ischemia-reperfusion injury patients: patients undergoing elective liver resection surgery with hepatic pedicle occlusion and reperfusion during the procedure.

Exclusion Criteria:

1) Patients with adverse events during surgery. 2) Patients in the end stage of disease with liver failure. 3) Liver tumor metastasis with concomitant severe heart failure or chronic renal insufficiency, etc. 4) Deemed unsuitable for participation in the study based on the judgment of the researchers.

-

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Criteria for liver ischemia-reperfusion injury patients: patients undergoing elective liver resection surgery with hepatic pedicle occlusion and reperfusion during the procedure.
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | 7days
  Length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China